CLINICAL TRIAL: NCT03589807
Title: A Phase II Study to Assess the Safety, Reactogenicity and Immunogenicity of Different Prime-Boost Vaccination Schedules of 2013 and 2017 A/H7N9 Inactivated Influenza Vaccines Administered Intramuscularly With or Without AS03 Adjuvant in Healthy Adults 19-50 Years of Age
Brief Title: 2013/2017 H7N9 Prime-Boost Interval
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 17-0078; HHSN272201300018I
Record Dates: First submitted 2018-06-28; First posted 2018-07-18 (Actual); Results first posted 2021-08-02 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2018-06-22

CONDITIONS: Avian Influenza; Influenza Immunisation
Keywords: A/H7N9; Adults; AS03; Immunogenicity; Influenza; Prime-Boost; Reactogenicity; Safety; Vaccine
MeSH Terms: conditions — Influenza in Birds; Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Heterologous Arm 1 (Experimental): 3.75 mcg per 0.5 ml dose of 2013 A/H7N9 Inactivated Influenza Virus Vaccine (IIV) + AS03 adjuvant administered intramuscularly on Day 1 and 3.75 mcg per 0.5 ml dose of 2017 A/H7N9 IIV + ASO3 adjuvant administered intramuscularly on Day 22. Phosphate buffered saline (PBS) diluent may be used to achieve targeted dosages. N=30
  Interventions: Biological: A/H7N9; Drug: AS03; Biological: Influenza Virus Vaccine, Monovalent A/H7N9 A/Shanghai/2/2013; Other: Phosphate Buffered Saline (PBS) diluent
- Heterologous Arm 2 (Experimental): 3.75 mcg per 0.5 ml dose of 2013 A/H7N9 IIV + AS03 adjuvant administered intramuscularly on Day 1 and 3.75 mcg per 0.5 ml dose of 2017 A/H7N9 IIV + ASO3 adjuvant administered intramuscularly on Day 121. PBS diluent may be used to achieve targeted dosages. N=30
  Interventions: Biological: A/H7N9; Drug: AS03; Biological: Influenza Virus Vaccine, Monovalent A/H7N9 A/Shanghai/2/2013; Other: Phosphate Buffered Saline (PBS) diluent
- Heterologous Arm 3 (Experimental): 3.75 mcg per 0.5 ml dose of 2013 A/H7N9 IIV + AS03 adjuvant administered intramuscularly on Day 1 and 15 mcg per 0.5 ml dose of 2017 A/H7N9 IIV administered intramuscularly on Day 121. PBS diluent may be used to achieve targeted dosages. N=30
  Interventions: Biological: A/H7N9; Drug: AS03; Biological: Influenza Virus Vaccine, Monovalent A/H7N9 A/Shanghai/2/2013; Other: Phosphate Buffered Saline (PBS) diluent
- Homologous Arm 1 (Experimental): 3.75 mcg per 0.5 ml dose of 2017 A/H7N9 IIV + AS03 adjuvant administered intramuscularly on Day 1 and Day 22. PBS diluent may be used to achieve targeted dosages. N=30
  Interventions: Biological: A/H7N9; Drug: AS03; Other: Phosphate Buffered Saline (PBS) diluent
- Homologous Arm 2 (Experimental): 3.75 mcg per 0.5 ml dose of 2017 A/H7N9 IIV + AS03 adjuvant administered intramuscularly on Day 1 and Day 121. PBS diluent may be used to achieve targeted dosages. N=30
  Interventions: Biological: A/H7N9; Drug: AS03; Other: Phosphate Buffered Saline (PBS) diluent
- Homologous Arm 3 (Experimental): 3.75 mcg per 0.5 ml dose of 2017 A/H7N9 IIV + AS03 Adjuvant administered intramuscularly on Day 1 and 15 mcg per 0.5 ml dose of 2017 A/H7N9 IIV administered intramuscularly on Day 121. PBS diluent may be used to achieve targeted dosages. N=30
  Interventions: Biological: A/H7N9; Drug: AS03; Other: Phosphate Buffered Saline (PBS) diluent

INTERVENTIONS:
Biological: A/H7N9 — Monovalent split 2017 A/H7N9 Inictivated Influenza Virus vaccine containing the HA and NA from low pathogenic avian influenza A/Hong Kong/125/2017 (H7N9) and the PB2, PB1, PA, NP, M and NS from A/Puerto Rico/8/1934 (H1N1).
Drug: AS03 — AS03 oil-in-water emulsion adjuvant.
Biological: Influenza Virus Vaccine, Monovalent A/H7N9 A/Shanghai/2/2013 — Monovalent split 2013 A/H7N9 Inavtivated Influenza Virus vaccine containing the HA and NA from avian influenza A/Shanghai/2/2013 (H7N9) and the PB2, PB1, PA, NP, M and NS from A/Puerto Rico/8/1934 (H1N1).
  Arms: Heterologous Arm 1; Heterologous Arm 2; Heterologous Arm 3
Other: Phosphate Buffered Saline (PBS) diluent — Diluent for Influenza Virus Vaccine.

SUMMARY:
This is a trial designed to assess the safety, reactogenicity and immunogenicity of one or two doses of monovalent inactivated split influenza 2013 and 2017 A/H7N9 virus vaccines administered intramuscularly at different dosages, given with or without AS03 adjuvant, using different vaccination schedules. This trial will enroll up to 180 males and non-pregnant females, 19 to 50 years of age, who are in good health and who are influenza A/H7 naïve. Subjects will be randomly assigned to 1 of 6 treatment arms (30 subjects per arm) to evaluate the interval between the first and second doses and the presence of the adjuvant in the first and second doses. The neuraminidase-specific antibody response and the neuraminidase content of the Inactivated Influenza Virus Vaccine will be determined using tests that are currently under development. Study duration is approximately 22 months with subject participation duration of approximately 18 months. The primary objectives of the study are: 1) to assess the safety and reactogenicity of 2013 and 2017 A/H7N9 IIVs given with or without AS03 adjuvant following receipt of each study vaccine; 2) to assess the serum hemagglutination inhibition (HAI) and neutralizing (Neut) antibody responses following receipt of the second study vaccine.

DETAILED DESCRIPTION:
This is a Phase II trial designed to assess the safety, reactogenicity and immunogenicity of one or two doses of monovalent inactivated split influenza 2013 and 2017 A/H7N9 virus vaccines (2013 and 2017 A/H7N9 IIVs) administered intramuscularly at different dosages (3.75 or 15 mcg of hemagglutinin (HA) per dose), given with or without AS03 adjuvant, using different heterologous and homologous prime-boost vaccination schedules. Phosphate buffered saline (PBS) diluent may be used to achieve targeted dosages. This trial will enroll up to 180 males and non-pregnant females, 19 to 50 years of age, inclusive, who are in good health and meet all eligibility criteria and who are influenza A/H7 vaccine/infection naïve by medical history. Subjects will be randomly assigned to 1 of 6 treatment arms (30 subjects per arm) evaluating the interval between the priming (first) and boosting (second) doses and the presence of the adjuvant in the priming (first) and boosting (second) doses. The neuraminidase-specific antibody response and the neuraminidase content of the Inactivated Influenza Virus Vaccine will be determined using tests that are currently under development. Study duration is approximately 22 months with subject participation duration of approximately 18 months. The primary objectives of the study are: 1) to assess the safety and reactogenicity of 2013 and 2017 A/H7N9 IIVs given with or without AS03 adjuvant following receipt of each study vaccine; 2) to assess the serum hemagglutination inhibition (HAI) and neutralizing (Neut) antibody responses following receipt of the second study vaccine. The secondary objectives are: 1) to assess unsolicited non-serious adverse events (AEs) following receipt of each study vaccine; 2) to assess medically-attended adverse events (MAAEs), including new-onset chronic medical conditions (NOCMCs) and potentially immune-mediated medical conditions (PIMMCs), following receipt of each study vaccine; 3) to assess the kinetics and durability of serum HAI and Neut antibody responses following receipt of each study vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent prior to initiation of any study procedures.
2. Are able to understand and comply with planned study procedures and be available for all study visits.
3. Must agree to the collection of venous blood per protocol.
4. Must agree to have residual specimens and samples/specimens collected during this trial specifically for the purpose of future research stored for future research use.
5. Are males or non-pregnant females, 19 to 50 years of age, inclusive.
6. Are in good health.

   * As determined by medical history and physical examination to evaluate acute or currently ongoing chronic medical diagnoses or conditions, defined as those that have been present for at least 90 days, which would affect the assessment of the safety of subjects or the immunogenicity of study vaccinations. Chronic medical diagnoses or conditions should be stable for the last 60 days (no hospitalizations, Emergency Room (ER), or urgent care for condition and no adverse symptoms that need medical intervention such as medication change/supplemental oxygen). This includes no change in chronic prescription medication, dose, or frequency as a result of deterioration of the chronic medical diagnosis or condition in the 60 days prior to enrollment. Any prescription change that is due to change of health care provider, insurance company, etc., or that is done for financial reasons, as long as in the same class of medication, will not be considered a deviation of this inclusion criterion. Any change in prescription medication due to improvement of a disease outcome, as determined by the site principal investigator or appropriate sub-investigator, will not be considered a deviation of this inclusion criterion. Subjects may be on chronic or as needed (prn) medications if, in the opinion of the site principal investigator or appropriate sub-investigator, they pose no additional risk to subject safety or assessment of reactogenicity and immunogenicity and do not indicate a worsening of medical diagnosis or condition. Similarly, medication changes subsequent to enrollment and study vaccination are acceptable provided there was no deterioration in the subject's chronic medical condition that necessitated a medication change, and there is no additional risk to the subject or interference with the evaluation of responses to study vaccination. Note: Topical, nasal, and inhaled medications (with the exception of inhaled corticosteroids as outlined in the Subject Exclusion Criteria), herbals, vitamins, and supplements are permitted.
7. Oral temperature is less than 100.0 degrees Fahrenheit.
8. Pulse is 47 to 100 beats per minute, inclusive.
9. Systolic blood pressure is 85 to 150 mmHg, inclusive.
10. Diastolic blood pressure is 55 to 95 mmHg, inclusive.
11. Erythrocyte Sedimentation Rate (ESR) is less than 30 mm per hour.
12. Women of childbearing potential must use an acceptable contraception method from 30 days before first study vaccination until 60 days after last study vaccination.

    - Not sterilized via tubal ligation, bilateral oophorectomy, salpingectomy, hysterectomy, or successful Essure(R) placement (permanent, non-surgical, non-hormonal sterilization) with documented radiological confirmation test at least 90 days after the procedure, and still menstruating or <1 year of the last menses if menopausal.

    -- Includes non-male sexual relationships, abstinence from sexual intercourse with a male partner, monogamous relationship with vasectomized partner who has been vasectomized for 180 days or more prior to the subject receiving the first study vaccination, barrier methods such as condoms or diaphragms with spermicide or foam, effective intrauterine devices, NuvaRing(R), and licensed hormonal methods such as implants, injectables, or oral contraceptives ("the pill").
13. Women of childbearing potential must have a negative urine or serum pregnancy test within 24 hours prior to study vaccination.

Exclusion Criteria:

1. Have an acute illness, as determined by the site principal investigator or appropriate sub-investigator, within 72 hours prior to study vaccination.

   * An acute illness which is nearly resolved with only minor residual symptoms remaining is allowable if, in the opinion of the site principal investigator or appropriate sub-investigator, the residual symptoms will not interfere with the ability to assess safety parameters as required by the protocol.
2. Have any medical disease or condition that, in the opinion of the site principal investigator or appropriate sub-investigator, is a contraindication to study participation.

   - Including acute or chronic medical disease or condition, defined as persisting for at least 90 days, that would place the subject at an unacceptable risk of injury, render the subject unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or the subject's successful completion of this trial.
3. Have immunosuppression as a result of an underlying illness or treatment, a recent history or current use of immunosuppressive or immunomodulating disease therapy.
4. Use of anticancer chemotherapy or radiation therapy (cytotoxic) within 3 years prior to study vaccination.
5. Have known active neoplastic disease or a history of any hematologic malignancy. Non-melanoma, treated, skin cancers are permitted.
6. Have known human immunodeficiency virus (HIV), hepatitis B, or hepatitis C infection.
7. Have known hypersensitivity or allergy to eggs, egg or chicken protein, squalene-based adjuvants, or other components of the study vaccine.
8. Have a history of severe reactions following previous immunization with licensed or unlicensed influenza vaccines.
9. Have a personal or family history of narcolepsy.
10. Have a history of Guillian-Barre Syndrome (GBS).
11. Have a history of convulsions or encephalomyelitis within 90 days prior to study vaccination.
12. Have a history of Potentially Immune-Mediated Medical Conditions (PIMMCs).
13. Have a history of alcohol or drug abuse within 5 years prior to study vaccination.
14. Have any diagnosis, current or past, of schizophrenia, bipolar disease, or other psychiatric diagnosis that may interfere with subject compliance or safety evaluations.

    - As determined by the site Principal Investigator or appropriate sub-investigator.
15. Have been hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others within 10 years prior to study vaccination.
16. Have taken oral or parenteral (including intra-articular) corticosteroids of any dose within 30 days prior to study vaccination.
17. Have taken high-dose inhaled corticosteroids within 30 days prior to each study vaccination.

    - High-dose defined as per age as using inhaled high-dose per reference chart in the National Heart, Lung and Blood Institute Guidelines for the Diagnosis and Management of Asthma (EPR-3) or other lists published in UPTODATE.
18. Received a licensed live vaccine within 30 days prior to the first study vaccination, or plan to receive a licensed live vaccine within 30 days before or after each study vaccination.
19. Received or plan to receive a licensed, inactivated vaccine (excluding all licensed, seasonal IIVs) within 14 days before or after each study vaccination.
20. Received or plan to receive a licensed, seasonal IIV within 21 days before or after each study vaccination
21. Received immunoglobulin or other blood products (except Rho D immunoglobulin) within 90 days prior to each study vaccination.
22. Received an experimental agent within 30 days prior to the first study vaccination, or expect to receive an experimental agent during the trial-reporting period.

    - Including vaccine, drug, biologic, device, blood product, or medication.

    -- Other than from participation in this trial.

    --- Approximately 12 months after the last study vaccination.
23. Are participating or plan to participate in another clinical trial with an interventional agent that will be received during the trial-reporting period.

    - Including licensed or unlicensed vaccine, drug, biologic, device, blood product, or medication.

    -- Approximately 12 months after the last study vaccination.
24. Received or plan to receive an influenza A/H7 vaccine or have a history of influenza A/H7 subtype infection.

    - And assigned to a treatment arm receiving influenza A/H7 vaccine, i.e., does not apply to documented placebo recipients.
25. Had substantial direct contact with live or freshly slaughtered poultry or pigeons while in mainland China within the past five years.

    - Substantial contact is defined as visited a poultry farm and/or a live poultry market.
26. Occupational exposure to or substantial direct physical contact with birds in the past year and through the 21 days after the last study vaccination.

    - Exposure to free range chickens in the yard is exclusionary. Casual contact with birds at petting zoos or county or state fairs, or having pet birds does not exclude subjects from study participation.
27. Female subjects who are breastfeeding or plan to breastfeed at any given time from the first study vaccination until 30 days after the last study vaccination.
28. Plan to travel outside the US (continental US, Hawaii, and Alaska) from the time of each study vaccination through 21 days after each study vaccination.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2018-08-21 (Actual); Primary Completion 2020-06-14 (Actual); Study Completion 2020-06-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Emory Children's Center - Pediatric Infectious Diseases, Atlanta, Georgia
  - Emory Vaccine Center - The Hope Clinic, Decatur, Georgia
  - University of Iowa - Vaccine Research and Education Unit, Iowa City, Iowa
  - Saint Louis University - Center for Vaccine Development, St Louis, Missouri
  - Duke Human Vaccine Institute - Duke Vaccine and Trials Unit, Durham, North Carolina
  - Baylor College of Medicine - Molecular Virology and Microbiology, Houston, Texas

REFERENCES:
- [Derived] El Sahly HM, Anderson EJ, Jackson LA, Neuzil KM, Atmar RL, Bernstein DI, Chen WH, Creech CB, Frey SE, Goepfert P, Meier J, Phadke V, Rouphael N, Rupp R, Stapleton JT, Spearman P, Walter EB, Winokur PL, Yildirim I, Williams TL, Oshinsky J, Coughlan L, Nijhuis H, Pasetti MF, Krammer F, Stadlbauer D, Nachbagauer R, Tsong R, Wegel A, Roberts PC. Anti-neuraminidase and anti-hemagglutinin stalk responses to different influenza a(H7N9) vaccine regimens. Vaccine. 2025 Feb 15;47:126689. doi: 10.1016/j.vaccine.2024.126689. Epub 2025 Jan 4. PMID 39756216
- [Derived] Rostad CA, Atmar RL, Walter EB, Frey S, Meier JL, Sherman AC, Lai L, Tsong R, Kao CM, Raabe V, El Sahly HM, Keitel WA, Whitaker JA, Smith MJ, Schmader KE, Swamy GK, Abate G, Winokur P, Buchanan W, Cross K, Wegel A, Xu Y, Yildirim I, Kamidani S, Rouphael N, Roberts PC, Mulligan MJ, Anderson EJ. A Phase 2 Clinical Trial to Evaluate the Safety, Reactogenicity, and Immunogenicity of Different Prime-Boost Vaccination Schedules of 2013 and 2017 A(H7N9) Inactivated Influenza Virus Vaccines Administered With and Without AS03 Adjuvant in Healthy US Adults. Clin Infect Dis. 2024 Jun 14;78(6):1757-1768. doi: 10.1093/cid/ciae173. PMID 38537255

RESULTS

PARTICIPANT FLOW:
Groups:
- 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22): 3.75 mcg per 0.5 ml dose of 2013 A/H7N9 Inactivated Influenza Virus Vaccine (IIV) + AS03 adjuvant administered intramuscularly on Day 1 and 3.75 mcg per 0.5 ml dose of 2017 A/H7N9 IIV + AS03 adjuvant administered intramuscularly on Day 22. Phosphate buffered saline (PBS) diluent may be used to achieve targeted dosages.
  A/H7N9: Monovalent split 2017 A/H7N9 Inactivated Influenza Virus vaccine containing the Hemagglutinin (HA) and Neuraminidase (NA) from low pathogenic avian influenza A/Hong Kong/125/2017 (H7N9) and other components from A/Puerto Rico/8/1934 (H1N1).
  AS03: Oil-in-water emulsion adjuvant.
  Influenza Virus Vaccine, Monovalent A/H7N9 A/Shanghai/2/2013: Monovalent split 2013 A/H7N9 Inactivated Influenza Virus vaccine containing the HA and NA from avian influenza A/Shanghai/2/2013 (H7N9) and other components from A/Puerto Rico/8/1934 (H1N1).
  Phosphate Buffered Saline (PBS) diluent: Diluent for Influenza Virus Vaccine.
- 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121): 3.75 mcg per 0.5 ml dose of 2013 A/H7N9 IIV + AS03 adjuvant administered intramuscularly on Day 1 and 3.75 mcg per 0.5 ml dose of 2017 A/H7N9 IIV + AS03 adjuvant administered intramuscularly on Day 121. PBS diluent may be used to achieve targeted dosages.
  A/H7N9: Monovalent split 2017 A/H7N9 Inactivated Influenza Virus vaccine containing the HA and NA from low pathogenic avian influenza A/Hong Kong/125/2017 (H7N9) and the PB2, PB1, PA, NP, M and NS from A/Puerto Rico/8/1934 (H1N1).
  AS03: Oil-in-water emulsion adjuvant.
  Influenza Virus Vaccine, Monovalent A/H7N9 A/Shanghai/2/2013: Monovalent split 2013 A/H7N9 Inactivated Influenza Virus vaccine containing the HA and NA from avian influenza A/Shanghai/2/2013 (H7N9) and other components from A/Puerto Rico/8/1934 (H1N1).
  Phosphate Buffered Saline (PBS) diluent: Diluent for Influenza Virus Vaccine.
- 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121): 3.75 mcg per 0.5 ml dose of 2013 A/H7N9 IIV + AS03 adjuvant administered intramuscularly on Day 1 and 15 mcg per 0.5 ml dose of 2017 A/H7N9 IIV administered intramuscularly on Day 121. PBS diluent may be used to achieve targeted dosages.
  A/H7N9: Monovalent split 2017 A/H7N9 Inactivated Influenza Virus vaccine containing the HA and NA from low pathogenic avian influenza A/Hong Kong/125/2017 (H7N9) and the PB2, PB1, PA, NP, M and NS from A/Puerto Rico/8/1934 (H1N1).
  AS03: Oil-in-water emulsion adjuvant.
  Influenza Virus Vaccine, Monovalent A/H7N9 A/Shanghai/2/2013: Monovalent split 2013 A/H7N9 Inactivated Influenza Virus vaccine containing the HA and NA from avian influenza A/Shanghai/2/2013 (H7N9) and other components from A/Puerto Rico/8/1934 (H1N1).
  Phosphate Buffered Saline (PBS) diluent: Diluent for Influenza Virus Vaccine.
- 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22): 3.75 mcg per 0.5 ml dose of 2017 A/H7N9 IIV + AS03 adjuvant administered intramuscularly on Day 1 and Day 22. PBS diluent may be used to achieve targeted dosages.
  A/H7N9: Monovalent split 2017 A/H7N9 Inactivated Influenza Virus vaccine containing the HA and NA from low pathogenic avian influenza A/Hong Kong/125/2017 (H7N9) and other components from A/Puerto Rico/8/1934 (H1N1).
  AS03: Oil-in-water emulsion adjuvant.
  Phosphate Buffered Saline (PBS) diluent: Diluent for Influenza Virus Vaccine.
- 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121): 3.75 mcg per 0.5 ml dose of 2017 A/H7N9 IIV + AS03 adjuvant administered intramuscularly on Day 1 and Day 121. PBS diluent may be used to achieve targeted dosages.
  A/H7N9: Monovalent split 2017 A/H7N9 Inactivated Influenza Virus vaccine containing the HA and NA from low pathogenic avian influenza A/Hong Kong/125/2017 (H7N9) and other components from A/Puerto Rico/8/1934 (H1N1).
  AS03: Oil-in-water emulsion adjuvant.
  Phosphate Buffered Saline (PBS) diluent: Diluent for Influenza Virus Vaccine.
- 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121): 3.75 mcg per 0.5 ml dose of 2017 A/H7N9 IIV + AS03 Adjuvant administered intramuscularly on Day 1 and 15 mcg per 0.5 ml dose of 2017 A/H7N9 IIV administered intramuscularly on Day 121. PBS diluent may be used to achieve targeted dosages.
  A/H7N9: Monovalent split 2017 A/H7N9 Inactivated Influenza Virus vaccine containing the HA and NA from low pathogenic avian influenza A/Hong Kong/125/2017 (H7N9) and other components from A/Puerto Rico/8/1934 (H1N1).
  AS03: Oil-in-water emulsion adjuvant.
  Phosphate Buffered Saline (PBS) diluent: Diluent for Influenza Virus Vaccine.
Period: Overall Study
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Started | 27 | 30 | 33 | 32 | 28 | 30
Completed | 27 | 23 | 31 | 28 | 26 | 29
Not Completed | 0 | 7 | 2 | 4 | 2 | 1
Not completed — Lost to Follow-up | 0 | 2 | 2 | 3 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 5 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Enrolled but treatment not administered | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population includes all participants who were enrolled in the study.
Groups:
- 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22): 3.75 mcg of 2013 A/H7N9 IIV+ AS03 adjuvant administered intramuscularly on Day 1 and 3.75 mcg of 2017 A/H7N9 IIV + AS03 adjuvant administered intramuscularly on Day 22.
- 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121): 3.75 mcg of 2013 A/H7N9 IIV + AS03 adjuvant administered intramuscularly on Day 1 and 3.75 mcg of 2017 A/H7N9 IIV + AS03 adjuvant administered intramuscularly on Day 121.
- 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121): 3.75 mcg of 2013 A/H7N9 IIV + AS03 adjuvant administered intramuscularly on Day 1 and 15 mcg of 2017 A/H7N9 IIV administered intramuscularly on Day 121.
- 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22): 3.75 mcg of 2017 A/H7N9 IIV + AS03 adjuvant administered intramuscularly on Day 1 and Day 22.
- 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121): 3.75 mcg of 2017 A/H7N9 IIV + AS03 adjuvant administered intramuscularly on Day 1 and Day 121.
- 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121): 3.75 mcg of 2017 A/H7N9 IIV + AS03 Adjuvant administered intramuscularly on Day 1 and 15 mcg of 2017 A/H7N9 IIV administered intramuscularly on Day 121.
- Total: Total of all reporting groups
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | Total
Number analyzed (Participants) | 27 | 30 | 33 | 32 | 28 | 30 | 180
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.3 (8.2) | 29.7 (7.5) | 29.6 (7.7) | 32.8 (9.2) | 31.2 (7.7) | 30.6 (8.4) | 31.0 (8.1)
Age, Customized [Number; unit: participants]
  19-34 | 16 | 24 | 25 | 19 | 19 | 19 | 122
  35-50 | 11 | 6 | 8 | 13 | 9 | 11 | 58
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 19 | 23 | 19 | 19 | 15 | 106
  Male | 16 | 11 | 10 | 13 | 9 | 15 | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 4 | 4 | 3 | 2 | 19
  Not Hispanic or Latino | 25 | 26 | 29 | 28 | 25 | 28 | 161
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 0 | 1 | 0 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 5 | 11 | 6 | 9 | 4 | 40
  White | 18 | 22 | 20 | 23 | 17 | 21 | 121
  More than one race | 3 | 0 | 2 | 2 | 2 | 2 | 11
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 27 | 30 | 33 | 32 | 28 | 30 | 180
Prior Seasonal Influenza Vaccination (Prior Seasons) [Count of Participants; unit: Participants]
  2016-2017 Reported | 15 | 16 | 14 | 20 | 19 | 17 | 101
  2016-2017 Not Reported | 12 | 14 | 19 | 12 | 9 | 13 | 79
  2017-2018 Reported | 17 | 18 | 22 | 20 | 20 | 18 | 115
  2017-2018 Not Reported | 10 | 12 | 11 | 12 | 8 | 12 | 65
Prior Seasonal Influenza Vaccination (Current Season) [Count of Participants; unit: Participants]
  2018-2019 Reported | 6 | 3 | 6 | 7 | 6 | 5 | 33
  2018-2019 Not Reported | 21 | 27 | 27 | 25 | 22 | 25 | 147
Prior Receipt of H5 Influenza Vaccine [Count of Participants; unit: Participants]
  No Prior H5 Influenza Vaccination(s) Reported | 24 | 29 | 30 | 31 | 27 | 28 | 169
  Reported Receipt of Prior H5 Influenza Vaccination(s) | 3 | 1 | 3 | 1 | 1 | 2 | 11
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: One subject in group 5 has missing value for BMI.
  kg/m^2
    number analyzed (Participants) | 27 | 30 | 33 | 32 | 27 | 30 | 179
    (all) | 27.07 (3.32) | 25.02 (4.27) | 28.32 (5.93) | 26.32 (4.96) | 27.17 (6.15) | 28.18 (6.80) | 27.02 (5.44)

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) of Serum Hemagglutinin Inhibition (HAI) Antibodies Against the Influenza A/H7N9 Study Vaccine Viruses on Day 43 in Participants Who Received Their Second Study Vaccination on Day 22.
Description: Blood was collected for HAI assay which was conducted with the 2017 H7N9 vaccine viruses as the antigens. Each sample was tested at least twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results at 21 days post second study vaccination (Day 43).
Time Frame: Day 43
Population: The modified intent-to-treat (mITT) population includes all participants who received study vaccination and contributed both pre- and at least one post-study vaccination venous blood samples for HAI antibody assays for which valid results were reported.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 27 | 0 | 0 | 31 | 0 | 0
titer
  A/Shanghai/2/2013 (A/H7N9) | 35.9 [22.5 to 57.5] |  |  | 19.5 [14.0 to 27.1] |  |
  A/Hong Kong/125/2017 (A/H7N9) | 75.7 [48.0 to 119.4] |  |  | 65.0 [42.4 to 99.5] |  |

2. Primary Outcome: Geometric Mean Titers (GMTs) of Serum Hemagglutinin Inhibition (HAI) Antibodies Against the Influenza A/H7N9 Study Vaccine Viruses on Day 142 in Participants Who Received Their Second Study Vaccination on Day 121.
Description: Blood was collected for HAI assay which was conducted with the 2017 H7N9 vaccine viruses as the antigens. Each sample was tested at least twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. The geometric mean titer was calculated for each study arm and stratum from the available results at 21 days post study vaccination (Day 142).
Time Frame: Day 142
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 0 | 22 | 31 | 0 | 26 | 27
titer
  A/Shanghai/2/2013 (A/H7N9) |  | 53.8 [31.7 to 91.4] | 22.6 [14.8 to 34.5] |  | 50.6 [30.8 to 83.2] | 17.0 [11.2 to 25.9]
  A/Hong Kong/125/2017 (A/H7N9) |  | 97.2 [55.9 to 169.0] | 43.1 [26.6 to 69.6] |  | 133.4 [83.6 to 212.6] | 33.2 [20.3 to 54.5]

3. Primary Outcome: Geometric Mean Titers (GMTs) of Serum Neutralizing (Neut) Antibodies Against the Influenza A/H7N9 Vaccine Viruses on Day 43 in Participants Who Received Their Second Study Vaccination on Day 22.
Description: Blood was collected for Neutralizing assay which was conducted with the H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results at 21 days post second study vaccination (Day 43).
Time Frame: Day 43
Population: The modified intent-to-treat (mITT) population includes all participants who received study vaccination and contributed both pre- and at least one post-study vaccination venous blood samples for Neut antibody assays for which valid results were reported.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 27 | 0 | 0 | 31 | 0 | 0
titer
  A/Shanghai/2/2013 (A/H7N9) | 86.4 [56.3 to 132.7] |  |  | 38.7 [27.8 to 53.9] |  |
  A/Hong Kong/125/2017 (A/H7N9) | 55.7 [37.7 to 82.1] |  |  | 51.2 [37.1 to 70.3] |  |

4. Primary Outcome: Geometric Mean Titers (GMTs) of Serum Neut Antibodies Against the Influenza A/H7N9 Study Vaccine Viruses on Day 142 in Participants Who Received Their Second Study Vaccination on Day 121
Description: Blood was collected for Neutralizing assay which was conducted with the H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results at 21 days post second study vaccination (Day 142).
Time Frame: Day 142
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 0 | 22 | 31 | 0 | 26 | 27
titer
  A/Shanghai/2/2013 (A/H7N9) |  | 286.6 [164.4 to 499.6] | 117.0 [70.7 to 193.6] |  | 178.0 [99.9 to 317.1] | 62.7 [38.0 to 103.5]
  A/Hong Kong/125/2017 (A/H7N9) |  | 146.1 [81.4 to 262.4] | 67.3 [42.2 to 107.4] |  | 202.0 [113.0 to 361.3] | 64.7 [40.3 to 103.9]

5. Primary Outcome: Number of Participants Reporting Serious Adverse Events (SAEs) From Day 1 Through Day 387 in Participants Who Received Their Second Study Vaccination on Day 22.
Description: SAEs included any untoward medical occurrence that resulted in death; was life threatening; was a persistent/significant disability/incapacity; required inpatient hospitalization or prolongation; or a congenital anomaly/birth defect.
Time Frame: Day 1 through Day 387
Population: The Safety Analysis population includes all participants who received study vaccination.
Measure: Count of Participants; unit: Participants
Groups:
- 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22): 3.75 mcg of 2013 A/H7N9 IIV + AS03 adjuvant administered intramuscularly on Day 1 and 3.75 mcg of 2017 A/H7N9 IIV + ASO3 adjuvant administered intramuscularly on Day 22.
- 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121): 3.75 mcg of 2013 A/H7N9 IIV + AS03 adjuvant administered intramuscularly on Day 1 and 3.75 mcg of 2017 A/H7N9 IIV + ASO3 adjuvant administered intramuscularly on Day 121.
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 27 | 0 | 0 | 32 | 0 | 0
Participants | 0 |  |  | 2 |  |

6. Primary Outcome: Number of Participants Reporting Serious Adverse Events (SAEs) From Day 1 Through Day 486 in Participants Who Received Their Second Study Vaccination on Day 121.
Description: as for outcome 5
Time Frame: Day 1 through Day 486
Population: The Safety Analysis population includes all participants who received study vaccination.
Measure: Count of Participants; unit: Participants
Groups:
- 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22): 3.75 mcg of 2013 A/H7N9 IIV + AS03 adjuvant administered intramuscularly on Day 1 and 3.75 mcg of 2017 A/H7N9 IIV + AS03 adjuvant administered intramuscularly on Day 22.
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 0 | 30 | 33 | 0 | 27 | 30
Participants |  | 0 | 1 |  | 0 | 1

7. Primary Outcome: Number of Participants Reporting Clinical Safety Laboratory Adverse Events (AEs) Post First Vaccination From Day 1 Through Day 8
Description: Laboratory parameters include alanine aminotransferase (ALT), bilirubin, creatinine, hemoglobin, platelets and white blood cells (WBC). Thresholds for adverse events were considered as ALT 44 IU/L or greater (female) or 61 IU/L or greater (male); bilirubin 1.30 mg/dL or greater; creatinine 1.1 mg/dL or greater (female) or 1.4 mg/dL or greater (male); hemoglobin 11.4 g/dL or lower (female) or 12.4 g/dL or lower (male); platelets 139 x10^3/µL or below or 416 x10^3/µL or greater; or WBC or 3.9 x10^3/µL or lower or 10.6 x10^3/µL or higher.
Time Frame: Day 1 through Day 8
Population: The Safety Analysis population includes all participants who received study vaccination. Participants with at least one lab result reported for Day 8 post first vaccination were included for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 27 | 30 | 33 | 31 | 27 | 29
Participants
  WBC | 3 | 4 | 1 | 0 | 2 | 1
  Hemoglobin | 2 | 3 | 2 | 1 | 1 | 2
  Platelets | 1 | 1 | 1 | 0 | 4 | 0
  ALT | 1 | 0 | 0 | 0 | 0 | 0
  Total Bilirubin | 0 | 1 | 0 | 0 | 0 | 1
  Creatinine | 1 | 0 | 1 | 0 | 1 | 0

8. Primary Outcome: Number of Participants Reporting Clinical Safety Laboratory Adverse Events (AEs) Post Second Vaccination From Day 121 Through Day 128 in Participants Who Received Their Second Study Vaccination on Day 121.
Description: as for outcome 7
Time Frame: Day 121 through Day 128
Population: The Safety Analysis population includes all participants who received study vaccination. Participants with at least one lab result reported for Day 8 post second vaccination were included for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 0 | 22 | 30 | 0 | 25 | 26
Participants
  WBC |  | 1 | 1 |  | 3 | 1
  Hemoglobin |  | 0 | 1 |  | 1 | 1
  Platelets |  | 0 | 0 |  | 1 | 0
  ALT |  | 0 | 0 |  | 0 | 1
  Total Bilirubin |  | 0 | 0 |  | 0 | 1
  Creatinine |  | 3 | 0 |  | 1 | 0

9. Primary Outcome: Number of Participants Reporting Clinical Safety Laboratory Adverse Events (AEs) Post Second Vaccination From Day 22 Through Day 29 in Participants Who Received Their Second Study Vaccination on Day 22.
Description: as for outcome 7
Time Frame: Day 22 through Day 29
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 26 | 0 | 0 | 29 | 0 | 0
Participants
  WBC | 4 |  |  | 0 |  |
  Hemoglobin | 1 |  |  | 3 |  |
  Platelets | 1 |  |  | 1 |  |
  ALT | 1 |  |  | 1 |  |
  Total Bilirubin | 0 |  |  | 0 |  |
  Creatine | 0 |  |  | 0 |  |

10. Primary Outcome: Number of Participants Reporting Solicited Injection Site Reactogenicity Events Post First Vaccination From Day 1 Through Day 8
Description: Injection site AEs solicited on a memory aid provided to participants included Pain, Tenderness, Itching/Pruritus, Ecchymosis/Bruising (functional grade based on interference with daily activities), Ecchymosis/Bruising (any measured value >0mm), Erythema/Redness (functional grade), Erythema/ Redness (any measured value >0mm), Induration/Swelling (functional grade), and Induration/Swelling (any measured value >0mm). Participants are considered reporting the injection site AE if they reported mild or greater severity at any time during the 8 days at or following the first vaccination.
Time Frame: Day 1 through Day 8
Population: The Safety Analysis population includes all participants who received study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 27 | 30 | 33 | 32 | 27 | 30
Participants | 25 | 27 | 30 | 28 | 26 | 29

11. Primary Outcome: Number of Participants Reporting Solicited Injection Site Reactogenicity Events Post Second Vaccination From Day 121 Through Day 128 in Participants Who Received Their Second Study Vaccination on Day 121.
Description: Injection site AEs solicited on a memory aid provided to participants included Pain, Tenderness, Itching/Pruritus, Ecchymosis/Bruising (functional grade based on interference with daily activities), Ecchymosis/Bruising (any measured value >0mm), Erythema/Redness (functional grade), Erythema/ Redness (any measured value >0mm), Induration/Swelling (functional grade), and Induration/Swelling (any measured value >0mm). Participants are considered reporting the injection site AE if they reported mild or greater severity at any time during the 8 days at or following the second vaccination.
Time Frame: Day 121 through Day 128
Population: The Safety Analysis population includes all participants who received study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 0 | 24 | 30 | 0 | 25 | 26
Participants |  | 23 | 12 |  | 24 | 10

12. Primary Outcome: Number of Participants Reporting Solicited Injection Site Reactogenicity Events Post Second Vaccination From Day 22 Through Day 29 in Participants Who Received Their Second Study Vaccination on Day 22.
Description: as for outcome 11
Time Frame: Day 22 through Day 29
Population: The Safety Analysis population includes all participants who received study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 26 | 0 | 0 | 31 | 0 | 0
Participants | 22 |  |  | 21 |  |

13. Primary Outcome: Number of Participants Reporting Solicited Systemic Reactogenicity Events Post First Vaccination From Day 1 Through Day 8
Description: Systemic AEs solicited on a memory aid provided to participants included Elevated Oral Temperature, Feverishness, Fatigue, Malaise, Myalgia, Arthralgia, Headache, and Nausea. Participants are considered reporting the systemic AE if they reported mild or greater severity at any time during the 8 days at or following the first vaccination.
Time Frame: Day 1 through Day 8
Population: The Safety Analysis population includes all participants who received study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 27 | 30 | 33 | 32 | 27 | 30
Participants | 17 | 12 | 18 | 10 | 17 | 16

14. Primary Outcome: Number of Participants Reporting Solicited Systemic Reactogenicity Events Post Second Vaccination From Day 121 Through Day 128 in Participants Who Received Their Second Study Vaccination on Day 121
Description: Systemic AEs solicited on a memory aid provided to participants included Elevated Oral Temperature, Feverishness, Fatigue, Malaise, Myalgia, Arthralgia, Headache, and Nausea. Participants are considered reporting the systemic AE if they reported mild or greater severity at any time during the 8 days at or following the second vaccination.
Time Frame: Day 121 through Day 128
Population: The Safety Analysis population includes all participants who received study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 0 | 24 | 30 | 0 | 25 | 26
Participants |  | 7 | 9 |  | 12 | 7

15. Primary Outcome: Number of Participants Reporting Solicited Systemic Reactogenicity Events Post Second Vaccination From Day 22 Through Day 29 in Participants Who Received Their Second Study Vaccination on Day 22.
Description: as for outcome 14
Time Frame: Day 22 through Day 29
Population: The Safety Analysis population includes all participants who received study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 26 | 0 | 0 | 31 | 0 | 0
Participants | 17 |  |  | 10 |  |

16. Primary Outcome: Percentage of Subjects Achieving Hemagglutination Inhibition (HAI) Antibody Titer of 1:40 or Greater Against the Influenza A/H7N9 Study Vaccine Viruses on Day 43 in Participants Who Received Their Second Study Vaccination on Day 22.
Description: Blood was collected for the HAI assay conducted with the H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The percentage of participants with HAI titer >= 1:40 was calculated for each study arm from the available results at 21 days post second study vaccination (Day 43).
Time Frame: Day 43
Population: The modified intent-to-treat (mITT) population includes all participants who received at least one study vaccination and contributed both pre- and at least one post-study vaccination venous blood samples for HAI antibody assays for which valid results were reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 27 | 0 | 0 | 31 | 0 | 0
percentage of participants
  A/Shanghai/2/2013 (A/H7N9) | 52 [32 to 71] |  |  | 35 [19 to 55] |  |
  A/Hong Kong/125/2017 (A/H7N9) | 81 [62 to 94] |  |  | 81 [63 to 93] |  |

17. Primary Outcome: Percentage of Subjects Achieving Hemagglutination Inhibition (HAI) Antibody Titer of 1:40 or Greater Against the Influenza A/H7N9 Study Vaccine Viruses on Day 142 in Participants Who Received Their Second Study Vaccination on Day 121.
Description: Blood was collected for the HAI assay conducted with the H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The percentage of participants with HAI titer >= 1:40 was calculated for each study arm from the available results at 21 days post second study vaccination (Day 142 ).
Time Frame: Day 142
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 0 | 22 | 31 | 0 | 26 | 27
percentage of participants
  A/Shanghai/2/2013 (A/H7N9) |  | 77 [55 to 92] | 32 [17 to 51] |  | 69 [48 to 86] | 19 [6 to 38]
  A/Hong Kong/125/2017 (A/H7N9) |  | 86 [65 to 97] | 61 [42 to 78] |  | 92 [75 to 99] | 59 [39 to 78]

18. Primary Outcome: Percentage of Participants Achieving Neutralizing (Neut) Antibody Titer of 1:40 or Greater Against the Influenza A/H7N9 Vaccine Viruses on Day 43 in Participants Who Received Their Second Study Vaccination on Day 22
Description: Blood was collected for the Neutralizing assay conducted with the H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The percentage of participants with Neut titer >= 1:40 was calculated for each study arm from the available results at 21 days post second study vaccination (Day 43).
Time Frame: Day 43
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 27 | 0 | 0 | 31 | 0 | 0
percentage of participants
  A/Shanghai/2/2013 (A/H7N9) | 85 [66 to 96] |  |  | 55 [36 to 73] |  |
  A/Hong Kong/125/2017 (A/H7N9) | 74 [54 to 89] |  |  | 74 [55 to 88] |  |

19. Primary Outcome: Percentage of Participants Achieving Neutralizing (Neut) Antibody Titer of 1:40 or Greater Against the Influenza A/H7N9 Vaccine Viruses on Day 142 in Participants Who Received Their Second Study Vaccination on Day 121.
Description: Blood was collected for the Neutralizing assay conducted with the H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The percentage of participants with Neut titer >= 1:40 was calculated for each study arm from the available results at 21 days post second study vaccination (Day 142).
Time Frame: Day 142
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 0 | 22 | 31 | 0 | 26 | 27
percentage of participants
  A/Shanghai/2/2013 (A/H7N9) |  | 95 [77 to 100] | 87 [70 to 96] |  | 92 [75 to 99] | 67 [46 to 83]
  A/Hong Kong/125/2017 (A/H7N9) |  | 91 [71 to 99] | 77 [59 to 90] |  | 92 [75 to 99] | 70 [50 to 86]

20. Primary Outcome: Percentage of Participants Achieving Hemagglutination Inhibition (HAI) Antibody Seroconversion Against the Influenza A/H7N9 Study Vaccine Viruses on Day 43 in Participants Who Received Their Second Study Vaccination on Day 22.
Description: Blood was collected for the HAI assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. Seroconversion was defined as HAI pre-vaccination titer <1:10 and post-vaccination titer >= 1:40 or pre-vaccination titer >= 1:10 and minimum 4-fold rise in post-vaccination antibody titer. 21 days after second study vaccination is Day 43.
Time Frame: Day 43
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 27 | 0 | 0 | 31 | 0 | 0
percentage of participants
  A/Shanghai/2/2013 (A/H7N9) | 52 [32 to 71] |  |  | 35 [19 to 55] |  |
  A/Hong Kong/125/2017 (A/H7N9) | 78 [58 to 91] |  |  | 81 [63 to 93] |  |

21. Primary Outcome: Percentage of Participants Achieving Hemagglutination Inhibition (HAI) Antibody Seroconversion Against the Influenza A/H7N9 Study Vaccine Viruses on Day 142 in Participants Who Received Their Second Study Vaccination on Day 121.
Description: Blood was collected for the HAI assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. Seroconversion was defined as HAI pre-vaccination titer <1:10 and post-vaccination titer >= 1:40 or pre-vaccination titer >= 1:10 and minimum 4-fold rise in post-vaccination antibody titer. 21 days after second study vaccination is Day 142.
Time Frame: Day 142
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 0 | 22 | 31 | 0 | 26 | 27
percentage of participants
  A/Shanghai/2/2013 (A/H7N9) |  | 77 [55 to 92] | 32 [17 to 51] |  | 69 [48 to 86] | 19 [6 to 38]
  A/Hong Kong/125/2017 (A/H7N9) |  | 86 [65 to 97] | 55 [36 to 73] |  | 85 [65 to 96] | 56 [35 to 75]

22. Primary Outcome: Percentage of Participants Achieving Neutralizing (Neut) Antibody Seroconversion Against the Influenza A/H7N9 Study Vaccine Viruses on Day 43 in Participants Who Received Their Second Study Vaccination on Day 22.
Description: Blood was collected for the Neutralizing assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. Seroconversion was defined as Neut pre-vaccination titer <1:10 and post-vaccination titer >= 1:40 or pre-vaccination titer >= 1:10 and minimum 4-fold rise in post-vaccination antibody titer. 21 days after second study vaccination is Day 43.
Time Frame: Day 43
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 27 | 0 | 0 | 31 | 0 | 0
percentage of participants
  Against A/Shanghai/2/2013 (A/H7N9) | 85 [66 to 96] |  |  | 55 [36 to 73] |  |
  A/Hong Kong/125/2017 (A/H7N9) | 74 [54 to 89] |  |  | 74 [55 to 88] |  |

23. Primary Outcome: Percentage of Participants Achieving Neutralizing (Neut) Antibody Seroconversion Against the Influenza A/H7N9 Study Vaccine Viruses on Day 142 in Participants Who Received Their Second Study Vaccination on Day 121.
Description: Blood was collected for the Neutralizing assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. Seroconversion was defined as Neut pre-vaccination titer <1:10 and post-vaccination titer >= 1:40 or pre-vaccination titer >= 1:10 and minimum 4-fold rise in post-vaccination antibody titer. 21 days after second study vaccination is Day 142.
Time Frame: Day 142
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 0 | 22 | 31 | 0 | 26 | 27
percentage of participants
  Against A/Shanghai/2/2013 (A/H7N9) |  | 95 [77 to 100] | 84 [66 to 95] |  | 92 [75 to 99] | 63 [42 to 81]
  A/Hong Kong/125/2017 (A/H7N9) |  | 91 [71 to 99] | 77 [59 to 90] |  | 92 [75 to 99] | 70 [50 to 86]

24. Secondary Outcome: Geometric Mean Titers (GMT) of Serum Hemagglutination Inhibition (HAI) Antibodies Against the Influenza A/H7N9 Study Vaccine Viruses on Day 1
Description: Blood was collected for HAI assay which was conducted with the 2013 and 2017 H7N9 vaccine viruses as the antigens. Each sample was tested at least twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results immediately prior to the first study vaccination (Day 1).
Time Frame: Day 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 27 | 28 | 33 | 31 | 27 | 30
titer
  A/Shanghai/2/2013 (A/H7N9) | 7.1 [NA to NA] — The limits of the 95% confidence interval were not calculable due to having a variance of 0. | 7.1 [NA to NA] — The limits of the 95% confidence interval were not calculable due to having a variance of 0. | 7.1 [NA to NA] — The limits of the 95% confidence interval were not calculable due to having a variance of 0. | 7.1 [NA to NA] — The limits of the 95% confidence interval were not calculable due to having a variance of 0. | 7.3 [7.0 to 7.6] | 7.1 [NA to NA] — The limits of the 95% confidence interval were not calculable due to having a variance of 0.
  A/Hong Kong/125/2017 (A/H7N9) | 7.4 [4.9 to 11.3] | 5.6 [4.7 to 6.8] | 6.8 [5.1 to 9.1] | 6.5 [5.0 to 8.4] | 6.0 [4.8 to 7.6] | 5.5 [4.5 to 6.9]

25. Secondary Outcome: Geometric Mean Titers (GMT) of Serum Hemagglutination Inhibition (HAI) Antibodies Against the Influenza A/H7N9 Study Vaccine Viruses on Day 22
Description: Blood was collected for HAI assay which was conducted with the 2013 and 2017 H7N9 vaccine viruses as the antigens. Each sample was tested at least twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results at 21 days post first study vaccination (Day 22).
Time Frame: Day 22
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 27 | 28 | 33 | 31 | 27 | 30
titer
  A/Shanghai/2/2013 (A/H7N9) | 8.8 [6.8 to 11.4] | 7.9 [6.9 to 9.0] | 7.6 [6.8 to 8.5] | 7.5 [7.0 to 8.1] | 7.1 [NA to NA] — The limits of the 95% confidence interval were not calculable due to having a variance of 0. | 7.1 [NA to NA] — The limits of the 95% confidence interval were not calculable due to having a variance of 0.
  A/Hong Kong/125/2017 (A/H7N9) | 9.7 [6.7 to 14.0] | 8.8 [5.9 to 12.9] | 8.2 [5.9 to 11.4] | 14.6 [8.8 to 24.2] | 8.9 [6.5 to 12.2] | 10.1 [6.5 to 15.5]

26. Secondary Outcome: Geometric Mean Titers (GMT) of Serum Hemagglutination Inhibition (HAI) Antibodies Against the Influenza A/H7N9 Study Vaccine Viruses on Day 202 in Participants Who Received Their Second Study Vaccination on Day 22
Description: Blood was collected for HAI assay which was conducted with the 2013 and 2017 H7N9 vaccine viruses as the antigens. Each sample was tested at least twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results at 180 days post second study vaccination (Day 202).
Time Frame: Day 202
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 27 | 0 | 0 | 30 | 0 | 0
titer
  A/Shanghai/2/2013 (A/H7N9) | 8.1 [6.9 to 9.4] |  |  | 7.4 [7.0 to 7.8] |  |
  A/Hong Kong/125/2017 (A/H7N9) | 24.7 [15.2 to 40.1] |  |  | 20.8 [13.5 to 32.1] |  |

27. Secondary Outcome: Geometric Mean Titers (GMT) of Serum Hemagglutination Inhibition (HAI) Antibodies Against the Influenza A/H7N9 Study Vaccine Viruses on Day 121 in Participants Who Received Their Second Study Vaccination on Day 121.
Description: Blood was collected for HAI assay which was conducted with the 2013 and 2017 H7N9 vaccine viruses as the antigens. Each sample was tested at least twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results immediately prior to second study vaccination (Day 121).
Time Frame: Day 121
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 0 | 25 | 32 | 0 | 27 | 28
titer
  A/Shanghai/2/2013 (A/H7N9) |  | 7.7 [6.6 to 8.8] | 7.1 [NA to NA] — The limits of the 95% confidence interval were not calculable due to having a variance of 0. |  | 7.1 [NA to NA] — The limits of the 95% confidence interval were not calculable due to having a variance of 0. | 7.1 [NA to NA] — The limits of the 95% confidence interval were not calculable due to having a variance of 0.
  A/Hong Kong/125/2017 (A/H7N9) |  | 9.3 [6.0 to 14.5] | 8.1 [6.0 to 10.9] |  | 9.8 [5.9 to 16.2] | 6.4 [4.8 to 8.5]

28. Secondary Outcome: Geometric Mean Titers (GMT) of Serum Hemagglutination Inhibition (HAI) Antibodies Against the Influenza A/H7N9 Study Vaccine Viruses on Day 301 in Participants Who Received Their Second Study Vaccination on Day 121
Description: Blood was collected for HAI assay which was conducted with the 2013 and 2017 H7N9 vaccine viruses as the antigens. Each sample was tested at least twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results at 180 days post second study vaccination (Day 301).
Time Frame: Day 301
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 0 | 20 | 27 | 0 | 25 | 25
titer
  A/Shanghai/2/2013 (A/H7N9) |  | 13.3 [9.5 to 18.6] | 8.8 [7.3 to 10.7] |  | 11.9 [8.8 to 16.0] | 7.1 [NA to NA] — The limits of the 95% confidence interval were not calculable due to having a variance of 0.
  A/Hong Kong/125/2017 (A/H7N9) |  | 47.3 [24.7 to 90.7] | 13.8 [8.6 to 22.0] |  | 38.8 [22.6 to 66.4] | 8.5 [6.4 to 11.1]

29. Secondary Outcome: Geometric Mean Titers (GMT) of Serum Neut Antibodies Against the Influenza A/H7N9 Study Vaccine Viruses on Day 1
Description: Blood was collected for Neut assay which was conducted with the 2013 and 2017 H7N9 vaccine viruses as the antigens. Each sample was tested at least twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results immediately prior to the first study vaccination (Day 1).
Time Frame: Day 1
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 27 | 28 | 33 | 31 | 27 | 30
titer
  A/Shanghai/2/2013 (A/H7N9) | 5.3 [4.9 to 5.9] | 5.4 [4.6 to 6.3] | 5.5 [4.6 to 6.5] | 5.1 [4.9 to 5.2] | 5.0 [NA to NA] — The limits of the 95% confidence interval were not calculable due to having a variance of 0. | 5.5 [4.6 to 6.7]
  A/Hong Kong/125/2017 (A/H7N9 | 5.3 [4.9 to 5.8] | 5.5 [4.7 to 6.4] | 5.3 [5.0 to 5.6] | 5.1 [4.9 to 5.4] | 5.2 [5.0 to 5.4] | 5.1 [4.9 to 5.4]

30. Secondary Outcome: Geometric Mean Titers (GMT) of Serum Neut Antibodies Against the Influenza A/H7N9 Study Vaccine Viruses on Day 22
Description: Blood was collected for Neut assay which was conducted with the 2013 and 2017 H7N9 vaccine viruses as the antigens. Each sample was tested at least twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results at 21 days post first study vaccination (Day 22).
Time Frame: Day 22
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 27 | 28 | 33 | 31 | 27 | 30
titer
  Against A/Shanghai/2/2013 (A/H7N9) | 11.5 [8.2 to 16.2] | 8.9 [7.2 to 11.0] | 9.6 [7.8 to 11.8] | 6.7 [5.7 to 7.8] | 6.6 [5.7 to 7.8] | 7.7 [6.2 to 9.5]
  A/Hong Kong/125/2017 (A/H7N9) | 8.1 [6.5 to 10.1] | 7.1 [6.0 to 8.4] | 7.5 [6.5 to 8.6] | 8.3 [6.8 to 10.0] | 8.6 [6.7 to 10.9] | 9.3 [7.4 to 11.7]

31. Secondary Outcome: Geometric Mean Titers (GMT) of Serum Neut Antibodies Against the Influenza A/H7N9 Study Vaccine Viruses on Day 202 in Participants Who Received Their Second Study Vaccination on Day 22
Description: Blood was collected for Neut assay which was conducted with the 2013 and 2017 H7N9 vaccine viruses as the antigens. Each sample was tested at least twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results at 180 days post second study vaccination (Day 202).
Time Frame: Day 202
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 27 | 0 | 0 | 30 | 0 | 0
titer
  A/Shanghai/2/2013 (A/H7N9) | 26.9 [20.7 to 34.8] |  |  | 13.3 [10.5 to 16.9] |  |
  A/Hong Kong/125/2017 (A/H7N9) | 18.5 [14.4 to 23.9] |  |  | 14.8 [12.1 to 18.1] |  |

32. Secondary Outcome: Geometric Mean Titers (GMT) of Serum Neut Antibodies Against the Influenza A/H7N9 Study Vaccine Viruses on Day 121 in Participants Who Received Their Second Study Vaccination on Day 121
Description: Blood was collected for Neut assay which was conducted with the 2013 and 2017 H7N9 vaccine viruses as the antigens. Each sample was tested at least twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results immediately prior to second study vaccination (Day 121).
Time Frame: Day 121
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 0 | 25 | 32 | 0 | 27 | 28
titer
  A/Shanghai/2/2013 (A/H7N9) |  | 13.9 [10.4 to 18.8] | 14.5 [11.4 to 18.4] |  | 8.5 [6.5 to 11.0] | 8.2 [6.8 to 9.9]
  A/Hong Kong/125/2017 (A/H7N9) |  | 11.2 [8.5 to 14.6] | 10.7 [8.7 to 13.1] |  | 9.9 [7.8 to 12.5] | 8.7 [7.3 to 10.5]

33. Secondary Outcome: Geometric Mean Titers (GMT) of Serum Neut Antibodies Against the Influenza A/H7N9 Study Vaccine Viruses on Day 301 in Participants Who Received Their Second Study Vaccination on Day 121
Description: Blood was collected for Neut assay which was conducted with the 2013 and 2017 H7N9 vaccine viruses as the antigens. Each sample was tested at least twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results at 180 days post second study vaccination (Day 301).
Time Frame: Day 301
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 0 | 20 | 27 | 0 | 25 | 25
titer
  A/Shanghai/2/2013 (A/H7N9) |  | 52.8 [29.9 to 93.2] | 27.9 [19.9 to 39.1] |  | 29.9 [19.2 to 46.6] | 14.9 [10.9 to 20.6]
  A/Hong Kong/125/2017 (A/H7N9) |  | 30.3 [18.7 to 49.0] | 17.8 [13.3 to 23.8] |  | 31.2 [20.2 to 48.1] | 15.8 [11.7 to 21.3]

34. Secondary Outcome: Number of Participants Who Received Their Second Study Vaccination on Day 22 Reporting Medically-Attended Adverse Events (MAAEs), New-Onset Chronic Medical Conditions (NOCMCs), and Potentially Immune-Mediated Medical Conditions (PIMMCs)
Description: Participants were queried at each visit for the occurrence of medically-attended adverse events (MAAEs), including new-onset chronic medical conditions (NOCMCs) and potentially immune-mediated medical conditions (PIMMCs) throughout the duration of the study.
Time Frame: Day 1 through Day 387
Population: The Safety Analysis population includes all participants who received study vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 27 | 0 | 0 | 32 | 0 | 0
Participants
  Medically-Attended Adverse Events | 9 |  |  | 8 |  |
  New Onset Chronic Medical Conditions | 0 |  |  | 1 |  |
  Potentially Immune-Mediated Medical Conditions | 0 |  |  | 0 |  |

35. Secondary Outcome: Number of Participants Who Received Their Second Study Vaccination on Day 121 Reporting Medically-Attended Adverse Events (MAAEs), New-Onset Chronic Medical Conditions (NOCMCs), and Potentially Immune-Mediated Medical Conditions (PIMMCs)
Description: as for outcome 34
Time Frame: Day 1 through Day 486
Population: The Safety Analysis population includes all participants who received study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 0 | 30 | 33 | 0 | 27 | 30
Participants
  Medically-Attended Adverse Events |  | 12 | 11 |  | 10 | 7
  New Onset Chronic Medical Conditions |  | 0 | 1 |  | 1 | 1
  Potentially Immune Mediated Medical Conditions |  | 0 | 0 |  | 0 | 0

36. Secondary Outcome: Number of Participants Reporting Unsolicited Non-serious AEs Post First Vaccination From Day 1 Through Day 22
Description: Adverse events were defined as any untoward medical occurrence in a participant administered a pharmaceutical product regardless of its causal relationship to the study treatment. Non-serious AEs were collected from participants at follow up visits through 21 days after the first study vaccination.
Time Frame: Day 1 through Day 22
Population: The Safety Analysis population includes all participants who received study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 27 | 30 | 33 | 32 | 27 | 30
Participants | 9 | 10 | 15 | 8 | 3 | 4

37. Secondary Outcome: Number of Participants Reporting Unsolicited Non-serious AEs Post Second Vaccination From Day 22 Through Day 43 in Participants Who Received Their Second Study Vaccination on Day 22
Description: Adverse events were defined as any untoward medical occurrence in a participant administered a pharmaceutical product regardless of its causal relationship to the study treatment. Non-serious AEs were collected from participants at follow up visits through 21 days after the second study vaccination.
Time Frame: Day 22 through Day 43
Population: The Safety Analysis population includes all participants who received study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 27 | 0 | 0 | 32 | 0 | 0
Participants | 7 |  |  | 4 |  |

38. Secondary Outcome: Number of Participants Reporting Unsolicited Non-serious AEs Post Second Vaccination From Day 121 Through Day 142 in Participants Who Received Their Second Study Vaccination on Day 121
Description: as for outcome 37
Time Frame: Day 121 through Day 142
Population: The Safety Analysis population includes all participants who received study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 0 | 30 | 33 | 0 | 27 | 30
Participants |  | 5 | 8 |  | 4 | 0

39. Secondary Outcome: Percentage of Participants Achieving Hemagglutination Inhibition (HAI) Antibody Seroconversion Against the Influenza A/H7N9 Study Vaccine Viruses on Day 22
Description: Blood was collected for HAI assay which was conducted with the 2013 and 2017 H7N9 vaccine viruses as the antigens. Each sample was tested at least twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. Seroconversion was defined as HAI pre-vaccination titer <1:10 and post-vaccination titer >= 1:40 or pre-vaccination titer >= 1:10 and minimum 4-fold rise in post-vaccination antibody titer. 21 days after first study vaccination is Day 22.
Time Frame: Day 22
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 27 | 28 | 33 | 31 | 27 | 30
percentage of participants
  A/Shanghai/2/2013 (A/H7N9) | 4 [0 to 19] | 4 [0 to 18] | 3 [0 to 16] | 0 [0 to 11] | 0 [0 to 13] | 0 [0 to 12]
  A/Hong Kong/125/2017 (A/H7N9) | 11 [2 to 19] | 11 [2 to 28] | 9 [2 to 24] | 26 [12 to 45] | 11 [2 to 29] | 17 [6 to 35]

40. Secondary Outcome: Percentage of Participants Achieving Hemagglutination Inhibition (HAI) Antibody Seroconversion Against the Influenza A/H7N9 Study Vaccine Viruses on Day 202 in Participants Who Received Their Second Study Vaccination on Day 22
Description: Blood was collected for HAI assay which was conducted with the 2013 and 2017 H7N9 vaccine viruses as the antigens. Each sample was tested at least twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. Seroconversion was defined as HAI pre-vaccination titer <1:10 and post-vaccination titer >= 1:40 or pre-vaccination titer >= 1:10 and minimum 4-fold rise in post-vaccination antibody titer. 180 days after second study vaccination is Day 202.
Time Frame: Day 202
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 27 | 0 | 0 | 30 | 0 | 0
percentage of participants
  A/Shanghai/2/2013 (A/H7N9) | 4 [0 to 19] |  |  | 0 [0 to 12] |  |
  A/Hong Kong/125/2017 (A/H7N9) | 41 [22 to 61] |  |  | 33 [17 to 53] |  |

41. Secondary Outcome: Percentage of Participants Achieving Hemagglutination Inhibition (HAI) Antibody Seroconversion Against the Influenza A/H7N9 Study Vaccine Viruses on Day 121 in Participants Who Received Their Second Study Vaccination on Day 121
Description: Blood was collected for HAI assay which was conducted with the 2013 and 2017 H7N9 vaccine viruses as the antigens. Each sample was tested at least twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. Seroconversion was defined as HAI pre-vaccination titer <1:10 and post-vaccination titer >= 1:40 or pre-vaccination titer >= 1:10 and minimum 4-fold rise in post-vaccination antibody titer. Immediately prior to second study vaccination is Day 121.
Time Frame: Day 121
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 0 | 25 | 32 | 0 | 27 | 28
percentage of participants
  A/Shanghai/2/2013 (A/H7N9) |  | 4 [0 to 20] | 0 [0 to 11] |  | 0 [0 to 13] | 0 [0 to 12]
  A/Hong Kong/125/2017 (A/H7N9) |  | 16 [5 to 36] | 6 [1 to 21] |  | 11 [2 to 29] | 7 [1 to 24]

42. Secondary Outcome: Percentage of Participants Achieving Hemagglutination Inhibition (HAI) Antibody Seroconversion Against the Influenza A/H7N9 Study Vaccine Virus on Day 301 in Participants Who Received Their Second Study Vaccination on Day 121
Description: Blood was collected for HAI assay which was conducted with the 2013 and 2017 H7N9 vaccine viruses as the antigens. Each sample was tested at least twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. Seroconversion was defined as HAI pre-vaccination titer <1:10 and post-vaccination titer >= 1:40 or pre-vaccination titer >= 1:10 and minimum 4-fold rise in post-vaccination antibody titer. 180 days after second study vaccination is Day 301.
Time Frame: Day 301
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 0 | 20 | 27 | 0 | 25 | 25
percentage of participants
  A/Shanghai/2/2013 (A/H7N9) |  | 10 [1 to 32] | 4 [0 to 19] |  | 12 [3 to 31] | 0 [0 to 14]
  A/Hong Kong/125/2017 (A/H7N9) |  | 75 [51 to 91] | 26 [11 to 46] |  | 56 [35 to 76] | 4 [0 to 20]

43. Secondary Outcome: Percentage of Participants Achieving Neutralizing (Neut) Antibody Seroconversion Against the Influenza A/H7N9 Study Vaccine Viruses on Day 22
Description: Blood was collected for Neutralizing assay which was conducted with the 2013 and 2017 H7N9 vaccine viruses as the antigens. Each sample was tested at least twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. Seroconversion was defined as Neut pre-vaccination titer <1:10 and post-vaccination titer >= 1:40 or pre-vaccination titer >= 1:10 and minimum 4-fold rise in post-vaccination antibody titer. 21 days after first study vaccination is Day 22.
Time Frame: Day 22
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 27 | 28 | 33 | 31 | 27 | 30
percentage of participants
  A/Shanghai/2/2013 (A/H7N9) | 11 [2 to 19] | 4 [0 to 18] | 3 [0 to 16] | 0 [0 to 11] | 0 [0 to 13] | 3 [0 to 17]
  A/Hong Kong/125/2017 (A/H7N9) | 4 [0 to 19] | 0 [0 to 12] | 0 [0 to 11] | 3 [0 to 17] | 7 [1 to 24] | 3 [0 to 17]

44. Secondary Outcome: Percentage of Participants Achieving Neutralizing (Neut) Antibody Seroconversion Against the Influenza A/H7N9 Study Vaccine Viruses on Day 202 in Participants Who Received Their Second Study Vaccination on Day 22
Description: Blood was collected for Neutralizing assay which was conducted with the 2013 and 2017 H7N9 vaccine viruses as the antigens. Each sample was tested at least twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. Seroconversion was defined as Neut pre-vaccination titer <1:10 and post-vaccination titer >= 1:40 or pre-vaccination titer >= 1:10 and minimum 4-fold rise in post-vaccination antibody titer. 180 days after second study vaccination is Day 202.
Time Frame: Day 202
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 27 | 0 | 00 | 30 | 0 | 0
percentage of participants
  A/Shanghai/2/2013 (A/H7N9) | 30 [14 to 50] |  |  | 10 [2 to 27] |  |
  A/Hong Kong/125/2017 (A/H7N9) | 19 [6 to 38] |  |  | 13 [4 to 31] |  |

45. Secondary Outcome: Percentage of Participants Achieving Neutralizing (Neut) Antibody Seroconversion Against the Influenza A/H7N9 Study Vaccine Viruses on Day 121 in Participants Who Received Their Second Study Vaccination on Day 121
Description: Blood was collected for Neutralizing assay which was conducted with the 2013 and 2017 H7N9 vaccine viruses as the antigens. Each sample was tested at least twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. Seroconversion was defined as Neut pre-vaccination titer <1:10 and post-vaccination titer >= 1:40 or pre-vaccination titer >= 1:10 and minimum 4-fold rise in post-vaccination antibody titer. Immediately prior to second study vaccination is Day 121.
Time Frame: Day 121
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 0 | 25 | 32 | 0 | 27 | 28
percentage of participants
  A/Shanghai/2/2013 (A/H7N9) |  | 12 [3 to 31] | 9 [2 to 25] |  | 4 [0 to 19] | 0 [0 to 12]
  A/Hong Kong/125/2017 (A/H7N9) |  | 4 [0 to 20] | 3 [0 to 16] |  | 4 [0 to 19] | 0 [0 to 12]

46. Secondary Outcome: Percentage of Participants Achieving Neutralizing (Neut) Antibody Seroconversion Against the Influenza A/H7N9 Study Vaccine Viruses on Day 301 in Participants Who Received Their Second Study Vaccination on Day 121
Description: Blood was collected for Neutralizing assay which was conducted with the 2013 and 2017 H7N9 vaccine viruses as the antigens. Each sample was tested at least twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. Seroconversion was defined as Neut pre-vaccination titer <1:10 and post-vaccination titer >= 1:40 or pre-vaccination titer >= 1:10 and minimum 4-fold rise in post-vaccination antibody titer. 180 days after second study vaccination is Day 301.
Time Frame: Day 301
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 0 | 20 | 27 | 0 | 25 | 25
percentage of participants
  A/Shanghai/2/2013 (A/H7N9) |  | 70 [46 to 88] | 44 [25 to 65] |  | 48 [28 to 69] | 20 [7 to 41]
  A/Hong Kong/125/2017 (A/H7N9) |  | 45 [23 to 68] | 22 [9 to 42] |  | 56 [35 to 76] | 16 [5 to 36]

47. Secondary Outcome: Percentage of Participants Achieving HAI Antibody Titer of 1:40 or Greater Against the Influenza A/H7N9 Study Vaccine Viruses on Day 1
Description: Blood was collected for HAI assay which was conducted with the 2013 and 2017 H7N9 vaccine viruses as the antigens. Each sample was tested at least twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. The percentage of participants with HAI titer >= 1:40 was calculated for each study arm from the available results immediately prior to the first study vaccination (Day 1).
Time Frame: Day 1
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 27 | 28 | 33 | 31 | 27 | 30
percentage of participants
  A/Shanghai/2/2013 (A/H7N9) | 0 [0 to 13] | 0 [0 to 12] | 0 [0 to 11] | 0 [0 to 11] | 0 [0 to 13] | 0 [0 to 12]
  A/Hong Kong/125/2017 (A/H7N9) | 11 [2 to 29] | 4 [0 to 18] | 6 [1 to 20] | 6 [1 to 21] | 4 [0 to 19] | 3 [0 to 17]

48. Secondary Outcome: Percentage of Participants Achieving HAI Antibody Titer of 1:40 or Greater Against the Influenza A/H7N9 Study Vaccine Viruses on Day 22
Description: Blood was collected for HAI assay which was conducted with the 2013 and 2017 H7N9 vaccine viruses as the antigens. Each sample was tested at least twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result The percentage of participants with HAI titer >= 1:40 was calculated for each study arm from the available results at 21 days post first study vaccination (Day 22).
Time Frame: Day 22
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 27 | 28 | 33 | 31 | 27 | 30
percentage of participants
  A/Shanghai/2/2013 (A/H7N9) | 4 [0 to 19] | 4 [0 to 18] | 3 [0 to 16] | 0 [0 to 11] | 0 [0 to 13] | 0 [0 to 12]
  A/Hong Kong/125/2017 (A/H7N9) | 15 [4 to 34] | 14 [4 to 33] | 12 [3 to 28] | 29 [14 to 48] | 11 [2 to 29] | 17 [6 to 35]

49. Secondary Outcome: Percentage of Participants Achieving HAI Antibody Titer of 1:40 or Greater Against the Influenza A/H7N9 Study Vaccine Viruses on Day 202 in Participants Who Received Their Second Study Vaccination on Day 22
Description: Blood was collected for HAI assay which was conducted with the 2013 and 2017 H7N9 vaccine viruses as the antigens. Each sample was tested at least twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. The percentage of participants with HAI titer >= 1:40 was calculated for each study arm from the available results at 180 days post first study vaccination (Day 202).
Time Frame: Day 202
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 27 | 0 | 0 | 30 | 0 | 0
percentage of participants
  A/Shanghai/2/2013 (A/H7N9) | 4 [0 to 19] |  |  | 0 [0 to 12] |  |
  A/Hong Kong/125/2017 (A/H7N9) | 48 [29 to 68] |  |  | 37 [20 to 56] |  |

50. Secondary Outcome: Percentage of Participants Achieving HAI Antibody Titer of 1:40 or Greater Against the Influenza A/H7N9 Study Vaccine Viruses on Day 121 in Participants Who Received Their Second Study Vaccination on Day 121
Description: Blood was collected for HAI assay which was conducted with the 2013 and 2017 H7N9 vaccine viruses as the antigens. Each sample was tested at least twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. The percentage of participants with HAI titer >= 1:40 was calculated for each study arm from the available results immediately prior to second study vaccination (Day 121).
Time Frame: Day 121
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 0 | 25 | 32 | 0 | 27 | 28
percentage of participants
  A/Shanghai/2/2013 (A/H7N9) |  | 4 [0 to 20] | 0 [0 to 11] |  | 0 [0 to 13] | 0 [0 to 12]
  A/Hong Kong/125/2017 (A/H7N9) |  | 20 [7 to 41] | 6 [1 to 21] |  | 11 [2 to 29] | 7 [1 to 24]

51. Secondary Outcome: Percentage of Participants Achieving HAI Antibody Titer of 1:40 or Greater Against the Influenza A/H7N9 Study Vaccine Viruses on Day 301 in Participants Who Received Their Second Study Vaccination on Day 121
Description: Blood was collected for HAI assay which was conducted with the 2013 and 2017 H7N9 vaccine viruses as the antigens. Each sample was tested at least twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. The percentage of participants with HAI titer >= 1:40 was calculated for each study arm from the available results at 180 days post first study vaccination (Day 301).
Time Frame: Day 301
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 0 | 20 | 27 | 0 | 25 | 25
percentage of participants
  A/Shanghai/2/2013 (A/H7N9) |  | 10 [1 to 32] | 4 [0 to 19] |  | 12 [3 to 31] | 0 [0 to 14]
  A/Hong Kong/125/2017 (A/H7N9) |  | 75 [51 to 91] | 30 [14 to 50] |  | 64 [43 to 82] | 4 [0 to 20]

52. Secondary Outcome: Percentage of Participants Achieving Neutralizing (Neut) Antibody Titer of 1:40 or Greater Against the Influenza A/H7N9 Vaccine Viruses on Day 1
Description: Blood was collected for Neutralizing assay which was conducted with the 2013 and 2017 H7N9 vaccine viruses as the antigens. Each sample was tested at least twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. The percentage of participants with Neut titer >= 1:40 was calculated for each study arm from the available results immediately prior to the first study vaccination (Day 1).
Time Frame: Day 1
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 27 | 28 | 33 | 31 | 27 | 30
percentage of participants
  A/Shanghai/2/2013 (A/H7N9) | 0 [0 to 13] | 4 [0 to 18] | 3 [0 to 16] | 0 [0 to 11] | 0 [0 to 13] | 3 [0 to 17]
  A/Hong Kong/125/2017 (A/H7N9) | 0 [0 to 13] | 4 [0 to 18] | 0 [0 to 11] | 0 [0 to 11] | 0 [0 to 13] | 0 [0 to 12]

53. Secondary Outcome: Percentage of Participants Achieving Neut Antibody Titer of 1:40 or Greater Against the Influenza A/H7N9 Study Vaccine Viruses on Day 22
Description: Blood was collected for Neut assay which was conducted with the 2013 and 2017 H7N9 vaccine viruses as the antigens. Each sample was tested at least twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result The percentage of participants with Neut titer >= 1:40 was calculated for each study arm from the available results at 21 days post first study vaccination (Day 22).
Time Frame: Day 22
Population: The modified intent-to-treat (mITT) population includes all participants who received at least one study vaccination and contributed both pre- and at least one post-study vaccination venous blood samples for Neut antibody assays for which valid results were reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 27 | 28 | 33 | 31 | 27 | 30
percentage of participants
  A/Shanghai/2/2013 (A/H7N9) | 11 [2 to 29] | 4 [0 to 18] | 3 [0 to 16] | 0 [0 to 11] | 0 [0 to 13] | 3 [0 to 17]
  A/Hong Kong/125/2017 (A/H7N9) | 4 [0 to 19] | 0 [0 to 12] | 0 [0 to 11] | 3 [0 to 17] | 7 [1 to 24] | 3 [0 to 17]

54. Secondary Outcome: Percentage of Participants Achieving Neut Antibody Titer of 1:40 or Greater Against the Influenza A/H7N9 Study Vaccine Viruses on Day 202 in Participants Who Received Their Second Study Vaccination on Day 22
Description: Blood was collected for Neut assay which was conducted with the 2013 and 2017 H7N9 vaccine viruses as the antigens. Each sample was tested at least twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. The percentage of participants with Neut titer >= 1:40 was calculated for each study arm from the available results at 180 days post first study vaccination (Day 202).
Time Frame: Day 202
Population: as for outcome 53
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 27 | 0 | 0 | 30 | 0 | 0
percentage of participants
  A/Shanghai/2/2013 (A/H7N9) | 33 [17 to 54] |  |  | 10 [2 to 27] |  |
  A/Hong Kong/125/2017 (A/H7N9) | 19 [6 to 38] |  |  | 13 [4 to 31] |  |

55. Secondary Outcome: Percentage of Participants Achieving Neut Antibody Titer of 1:40 or Greater Against the Influenza A/H7N9 Study Vaccine Viruses on Day 121 in Participants Who Received Their Second Study Vaccination on Day 121
Description: Blood was collected for NEUT assay which was conducted with the 2013 and 2017 H7N9 vaccine viruses as the antigens. Each sample was tested at least twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. The percentage of participants with Neut titer >= 1:40 was calculated for each study arm from the available results immediately prior to second study vaccination (Day 121).
Time Frame: Day 121
Population: as for outcome 53
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 0 | 25 | 32 | 0 | 27 | 28
percentage of participants
  A/Shanghai/2/2013 (A/H7N9) |  | 12 [3 to 31] | 9 [2 to 25] |  | 4 [0 to 19] | 0 [0 to 12]
  A/Hong Kong/125/2017 (A/H7N9) |  | 4 [0 to 20] | 3 [0 to 16] |  | 4 [0 to 19] | 0 [0 to 12]

56. Secondary Outcome: Percentage of Participants Achieving Neut Antibody Titer of 1:40 or Greater Against the Influenza A/H7N9 Study Vaccine Viruses on Day 301 in Participants Who Received Their Second Study Vaccination on Day 121
Description: Blood was collected for Neut assay which was conducted with the 2013 and 2017 H7N9 vaccine viruses as the antigens. Each sample was tested at least twice per antigen per the laboratory's standard operating procedure, and the geometric mean of the replicate results of each antigen was calculated as that sample's result. The percentage of participants with Neut titer >= 1:40 was calculated for each study arm from the available results at 180 days post second study vaccination (Day 301).
Time Frame: Day 301
Population: as for outcome 53
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
Number analyzed (Participants) | 0 | 20 | 27 | 0 | 25 | 25
percentage of participants
  A/Shanghai/2/2013 (A/H7N9) |  | 70 [46 to 88] | 44 [25 to 65] |  | 48 [28 to 69] | 20 [7 to 41]
  A/Hong Kong/125/2017 (A/H7N9) |  | 45 [23 to 68] | 22 [9 to 42] |  | 56 [35 to 76] | 16 [5 to 36]

ADVERSE EVENTS:
Time Frame: Solicited events were collected from the time of each vaccination through 7 days after each vaccination. Unsolicited non-serious AEs were collected from the time of each vaccination through about 21 days after each vaccination. SAEs and MAAEs, including NOCMCs and PIMMCs, were collected from the time of first vaccination through the final study visit, about 12 months after the last vaccination, totaling 13 or 16 months for those who received the second vaccine on day 21 or day 121, respectively.
Description: Number of subjects at risk represent the number of subjects who received at least one study vaccination.
Arm/Group | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121)
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/30 | 0/33 | 0/32 | 0/27 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/30 | 1/33 | 2/32 | 0/27 | 1/30
Other Adverse Events (participants affected / at risk) | 27/27 | 30/30 | 33/33 | 31/32 | 27/27 | 29/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) (N=27) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) (N=30) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) (N=33) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) (N=32) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) (N=27) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) (N=30)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Organ donor (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) (N=27) | 2013 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) (N=30) | 2013 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) (N=33) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D22) (N=32) | 2017 3.75 A/H7N9+AS03| 2017 3.75 A/H7N9 + AS03 (D1-D121) (N=27) | 2017 3.75 A/H7N9+AS03| 2017 15 A/H7N9 (D1-D121) (N=30)
Nuasea (Gastrointestinal disorders) | 2 (2) | 3 (4) | 6 (7) | 4 (5) | 6 (6) | 1 (1)
Fatigue (General disorders) | 14 (21) | 9 (13) | 11 (15) | 13 (18) | 9 (12) | 14 (19)
Feeling hot (General disorders) | 4 (4) | 6 (7) | 3 (3) | 4 (5) | 6 (6) | 2 (2)
Injection site erythema (General disorders) | 4 (4) | 9 (10) | 11 (12) | 12 (15) | 15 (16) | 11 (15)
Injection site haemorrhage (General disorders) | 1 (2) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 3 (3)
Injection site induration (General disorders) | 4 (5) | 10 (12) | 9 (9) | 8 (12) | 13 (19) | 5 (5)
Injection site pain (General disorders) | 17 (27) | 21 (31) | 15 (18) | 16 (23) | 17 (27) | 15 (17)
Injection site pain (tenderness) (General disorders) | 23 (43) | 28 (49) | 27 (33) | 24 (41) | 26 (47) | 28 (32)
Injection site pruritus (General disorders) | 2 (2) | 3 (3) | 4 (4) | 2 (2) | 5 (6) | 2 (2)
Malaise (General disorders) | 7 (9) | 5 (8) | 4 (5) | 6 (8) | 8 (9) | 5 (6)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (3) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3) | 4 (5) | 3 (3) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 1 (3) | 0 (0)
Blood pressure diastolic increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 1 (1) | 0 (0)
Hemoglobin decreased (Investigations) | 3 (6) | 3 (3) | 3 (5) | 4 (9) | 1 (2) | 2 (4)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Platelet count increased (Investigations) | 1 (3) | 1 (2) | 1 (2) | 1 (1) | 2 (4) | 0 (0)
White blood cell count decreased (Investigations) | 3 (7) | 4 (7) | 2 (3) | 0 (0) | 6 (9) | 1 (2)
White blood cell count increased (Investigations) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 5 (7) | 3 (3) | 4 (4) | 3 (4) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 12 (18) | 10 (12) | 12 (12) | 8 (11) | 11 (14) | 11 (11)
Headache (Nervous system disorders) | 9 (9) | 6 (8) | 11 (12) | 8 (10) | 10 (13) | 6 (7)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (4) | 1 (1) | 2 (2) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-12-18): https://cdn.clinicaltrials.gov/large-docs/07/NCT03589807/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-18): https://cdn.clinicaltrials.gov/large-docs/07/NCT03589807/SAP_001.pdf